CLINICAL TRIAL: NCT05048368
Title: A Pharmacokinetic Study of Larotinib in Subjects With Mild/Moderate Hepatic Impairment and in Healthy Subjects With Normal Hepatic Function
Brief Title: Pharmacokinetics Study of Larotinib in Subjects With Impaired Hepatic Function
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z650-HI-105
Record Dates: First submitted 2021-09-06; First posted 2021-09-17 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer; Advanced Solid Tumor
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is divided into four cohorts: healthy subjects in cohort A and C, mild liver function impairment subjects in cohort B, and moderateliver function impairment subjects in cohort D. Cohorts A and B, C and D should be matched in terms of gender, age, and body mass index (BMI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A-Larotinib (Experimental): Cohort A:Healthy participants with normal hepatic function （match to subjects with mild hepatic impairment_cohort B）
  Interventions: Drug: Larotinib
- Cohort B-Larotinib (Experimental): Subjects with mild hepatic impairment
  Interventions: Drug: Larotinib
- Cohort C-Larotinib (Experimental): Healthy participants with normal hepatic function （match to subjects with moderate hepatic impairment_cohort D）
  Interventions: Drug: Larotinib
- Cohort D-Larotinib (Experimental): Subjects with moderate hepatic impairment.
  Interventions: Drug: Larotinib

INTERVENTIONS:
Drug: Larotinib — Capsules, Oral, 350 mg, single dose, one day

SUMMARY:
To evaluate the pharmacokinetics and safety of Larotinib in subjects with mild and moderate hepatic function impairment and healthy subjects in a single-center, non-randomized, open, single-dose administration

DETAILED DESCRIPTION:
A phase I, a single-center, non-randomized, open, single-dose administration study to explore the safety, pharmacokinetics of Larotinib in subjects with mild and moderate hepatic function impairment and healthy subjects with normal hepatic function.

This study is divided into four cohorts, cohort A and cohort C in healthy subjects, cohort B for mild hepatic function impairment participants, cohort D for moderate hepatic function impairment, participants in cohort A and cohort B, group C and group D should be matched in terms of sex, age, and body mass index (BMI). A total of 32 subjects, 8 in each cohort, both male and female, are planned to be enrolled. If a complete PK blood sample is not collected due to subjects' early withdrawal from the study, new subjects will be enrolled to meet the pharmacokinetic parameters that can be evaluated for each cohort of 8 subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects with normal hepatic function (cohorts A and C) :
* 1. Sign the informed consent form before the trial；
* 2. subjects and must be 18 to 70 years of age inclusive, Male or female. body weight >50 kg (male) or ≥45 kg (female) at screening. (BMI) : 18-30 kg/m^2, (including critical value) [BMI= weight (kg)/height^2 (m^2)] (BMI matching ±15% with liver dysfunction cohort);
* 3.Must be in good health as determined by past medical history, physical examination, vital signs, ECG, and laboratory tests at Screening；
* 4.Subjects (including partners) have no pregnancy plan within 6 months after the last dose of study drug and voluntarily take effective contraceptive measures.
* Subjects with mild/ Moderate hepatic Impairment (cohorts B and D) :
* 1. Sign the informed consent form before the trial.
* 2. subjects and must be 18 to 70 years of age inclusive, Male or female. body weight >50 kg (male) or ≥45 kg (female) at screening. (BMI) : 18-30 kg/m^2；
* 3. Must satisfy the criteria for hepatic Impairment as evidenced by a Child-Pugh class of A or B at Screening:Class A; Mild; Child-Pugh score 5-6；Class B; Moderate; Child-Pugh score 7-9
* 4. The liver function status of the subjects was determined to be stable between 1 month before taking the experimental drug and the end of the study, with no significant change.
* 5. Subjects (including partners) have no pregnancy plan within 6 months after the last dose of study drug and voluntarily take effective contraceptive measures.

Exclusion Criteria:

* ALL subjects
* 1. The subject has been diagnosed with acquired immune deficiency syndrome (AIDS), or tests positive for human immunodeficiency virus (HIV).
* 2. Currently suffering from any bleeding disease, such as gastric and duodenal ulcer
* 3. Those who had undergone major surgery within 6 months before the screening period or the surgical incision did not completely heal;
* 4. History of hand foot syndrome;
* 5. Those who have a history of liver cancer or other malignant tumors before signing the informed consent
* 6. Those who have a history of gastrointestinal and renal diseases or surgery that may affect drug absorption, distribution, metabolism and excretion within 6 months before screening, or have diseases that can reduce compliance
* 7. Take any food or beverage products containing alcohol, caffeine, xanthine and grapefruit within 48 hours prior to the first dose.
* 8. The subject has received blood within 1 month, or donated loss of blood over 400 mL within 3 months prior to the screening
* 9. Have a history of alcoholism or positive alcohol breath test during the screening period;
* 10. Those who smoke more than 5 cigarettes a day or habitually use nicotine containing products 3 months before screening
* 11. Those who had a history of drug abuse or used drugs within 2 years before screening or those who were positive for urinary drug screening during the screening period Allergic constitution
* 12. Allergic constitution
* 13. Within 28 days before screening, inhibitors or inducers of CYP3A4, cyp2c8, CYP2C19 and P-gp were used
* 14. Participated in any other intervention clinical trial within 3 months before screening
* 15. Female subjects with positive pregnancy test results or breastfeeding during screening;
* 16. Any other circumstances that the investigator considers unsuitable for participation in this study
* The following exclusion criteria apply only to healthy subjects with normal hepatic function (cohorts A and C) :
* 17. he subject has evidence of clinically significant cardiovascular, GI, renal, respiratory, endocrine, hematological, neurological, or psychiatric disease or abnormalities.
* 18. The subject tests positive for HBsAg or Hepatitis C antibody
* 19. The subject has used any prescription or nonprescription drugs within 2 weeks prior to the screening.
* The following exclusion criteria apply only to subjects with mild/ Moderate hepatic Impairment (cohorts B and D) :
* 17. The following exclusion criteria apply only to subjects with liver function impairment (cohorts B and D) :
* a) ALT>10×ULN；
* b) AST> 10×ULN；
* c) Absolute count of neutrophils <0.75×10^9/L;
* d) PLT<50×10^9/L
* e) HGB<60 g/L
* f) AFP >100 ng/mL; If 20 ng/mL≤AFP≤100 ng/mL, liver MRI are required to exclude subjects with suspected HCC.
* g) eGFR<60 mL/min/1.73m^2.
* h) Male：QTcF> 450 msec，Female：QTcF>470 msec。
* 18. The subject has any of the following conditions: Diseases affecting bile excretion such as biliary obstruction; Drug induced liver injury; History of liver transplantation; Liver failure, or liver cirrhosis patients with complications such as hepatic encephalopathy, rupture and bleeding of esophageal and gastric varices, etc; Patients with severe or advanced peritoneal effusion or pleural effusion need puncture drainage and albumin supplementation. Patients with hepatorenal syndrome.
* 19. Previous severe esophagogastric varices or previous portosystemic shunt, including transjugular intrahepatic portosystemic shunt (TIPS)
* 20. Cardiovascular events occurred within 6 months before screening
* 21. Those who use prescription drugs, over-the-counter drugs, Chinese herbal medicine or food supplements other than drugs for the treatment of liver function impairment and other accompanying diseases within 14 days before screening;
* 22. Medical conditions which are not adequately and stably controlled on stable doses of medications or which, in the clinical opinion of the Principal Investigator, may interfere with study procedures or participant safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-10-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day 1 to Day 7
  Maximum plasma concentration of study drugs
Area Under Curve From 0 to Infinity (AUC0-infinity) | Day 1 to Day 7
  AUC0-infinity represents the area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity

SECONDARY OUTCOMES:
Adverse Event | Day-7 to Day 14
  New abnormal findings or worsening of baseline conditions were reported as Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Miao, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China